CLINICAL TRIAL: NCT03581448
Title: Virtual Neuroprosthesis: Restoring Autonomy to People Suffering From Neurotrauma
Brief Title: Virtual Neuroprosthesis: Restoring a Sense of Touch to Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Collaborators: University of Utah (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FloridaAU; R01EB025819 (NIH)
Record Dates: First submitted 2018-06-13; First posted 2018-07-10 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Amputation

STUDY DESIGN:
Intervention Model Description: Study falls under device feasibility: An intervention of a device product is being evaluated in a small clinical trial to determine the feasibility of the product; or a clinical trial to test a prototype device for feasibility and not health outcomes. Such studies are conducted to confirm the design and operating specifications of a device before beginning a full clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nerve Growth During Prosthesis Control (Experimental): Determine the optimum conditions that promote sensory restoration in limb-absent people, with an adaptive haptic feedback control law that mimics the experience of neural plasticity.
  The intervention Sensory Restoration During Prosthesis Control will be used.
  Interventions: Behavioral: Sensory Restoration During Prosthesis Control

INTERVENTIONS:
Behavioral: Sensory Restoration During Prosthesis Control — Human subjects who use a robotic arm/hand interface will experience variable sensations of touch over time.

SUMMARY:
The overall goal of this project is to develop a virtual neuroprosthesis in which a facsimile of a neural implant is externalized and housed in a well-controlled microfluidic chamber, thereby abating the intrinsic limitations of highly invasive studies with neural implants. Able-bodied and upper limb amputee subjects will be recruited to control a dexterous artificial hand and arm with electromyogram signals while electroencephalogram (EEG) signals are simultaneously measured. Robotic grip force measurements will be biomimetically converted into electrical pulses similar to those found in the peripheral nervous system to catalyze in vitro nerve regeneration after neurotrauma. The synergistic contributions of this multidisciplinary project will lead to a transformative understanding of the symbiotic interaction of neural plasticity within human-robotic systems. Currently, there is no systematic understanding of how tactile feedback signals can contribute to the neural regeneration of afferent neural pathways to restore somatosensation and improve motor function in amputees fitted with neuroprosthetic limbs. Tackling this problem will be a significant breakthrough for the important field of neuroprosthetics.

DETAILED DESCRIPTION:
Over one week, neurobehavioral processes will be examined in people controlling a robotic arm and hand to perform simple motor tasks (e.g. fragile object transportation), while a virtual peripheral nerve regeneration protocol provides users with biologically-realistic, idiosyncratic parameters for the restoration of haptic sensation (in double-blind fashion, the cellular neurophysiologists characterizing neural regeneration with microscopy are unaware of subjects' name and condition; and the human-subject experimenters are unaware of the haptic feedback parameter that will be used in the experiment each day, which is entered by the neurophysiologist in a black-box section of the software in the case of microscopic evaluation of nerve regeneration (early part of the project), or which is automatically input by the system in the case of real time impedimetric measurements (later part of the project)).

The main experimental factors are 'haptic feedback', with three modalities: full, partial (nerve-regeneration dependent) and null; and to challenge human control strategy and impose demand on haptic information, the 'transported object weight' (heavy, medium and lightweight).

Recording techniques: Subjects' electroencephalography (EEG), electromyography (EMG) and behavioral performance.

ELIGIBILITY:
Inclusion Criteria:

* No neurological impairment of tactile sensation.

Exclusion Criteria:

* Younger than 18 or older than 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Engeberg, Ph.D., Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Gender, ethnicity (if voluntarily disclosed), and nature of upper-limb absence (If applicable) are recorded. This information is reported in corresponding journal and conference publications.
Supporting Information: Study Protocol, SAP
Time Frame: Within 1 year after primary completion.
Access Criteria: Open access.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Exclusion criteria preventing subjects from participating are an amputation wound that has not yet healed, the absence of a suitable length of residual limb for placement of haptic feedback controller and EMG sensors, presence of pain that prevents utilization of those experimental appliances and the use of psychoactive drugs that modifies baseline neural activity.
Groups:
- Experimental: Nerve Growth During Prosthesis Control: Determine the optimum conditions that promote sensory restoration in limb-absent people, with an adaptive haptic feedback control law that mimics the experience of neural plasticity.
  The intervention Sensory Restoration During Prosthesis Control will be used.
Period: Overall Study
Arm/Group | Experimental: Nerve Growth During Prosthesis Control
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Amputees
Groups:
- Nerve Growth During Prosthesis Control: Determine the optimum conditions that promote sensory restoration in limb-absent people, with an adaptive haptic feedback control law that mimics the experience of neural plasticity.
  The intervention Sensory Restoration During Prosthesis Control will be used.
  Sensory Restoration During Prosthesis Control: Human subjects who use a robotic arm/hand interface will experience variable sensations of touch over time.
Arm/Group | Nerve Growth During Prosthesis Control
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Artificial Hand Grasp Performance Metrics
Description: The percentage that grasped objects are successfully transported without slip or drop when controlled by amputees using an artificial hand.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: percentage of successful transportation
Arm/Group | Experimental: Nerve Growth During Prosthesis Control
Number analyzed (Participants) | 21
percentage of successful transportation | 90.6 (14.0)

2. Secondary Outcome: Dorsal Root Ganglia Neurite Regeneration
Description: The length of neurite regeneration 1 week post-axotomy will be quantified. The dorsal root ganglia will be cultured in vitro in a multichannel microelectrode array. The neural culture will be electrically stimulated based on the touch sensations from the artificial hand that is used by amputees. The fingertip touch sensations will be biomimetically converted into pulses that resemble action potentials for the electrical stimulation. The length of neurite regeneration was quantified using NeuronJ to compare images at the beginning and endpoints of the study.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Experimental: Nerve Growth During Prosthesis Control
Number analyzed (Participants) | 21
micrometer | 2309 (222)

ADVERSE EVENTS:
Time Frame: 1 week
Description: Application of electroencephalogram electrodes and arm sensors present a small risk of skin irritation that is extremely rare and usually disappears within a day or two. There are small risks of tension or fatigue in the muscles; of visual fatigue while concentrating on the computer screen or robotic hand.
Arm/Group | Experimental: Nerve Growth During Prosthesis Control
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT03581448/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT03581448/ICF_001.pdf